CLINICAL TRIAL: NCT06543160
Title: Immediate Skin-to-Skin Contact and Breastfeeding During Caesarean Section: A Randomized Controlled Trial on Early Neonatal Hypoglycemia in Late Preterm and Term Infants
Brief Title: Immediate Skin-To-Skin Contact and Early Breastfeeding During Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qingdao Municipal Hospital (Other)
Responsible Party: Principal Investigator, Jia Qiao, RN, Qingdao Municipal Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Grant No.(2023LinShenZi No.123
Record Dates: First submitted 2024-07-31; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Hypoglycemia
Keywords: neonatal hypoglycemia; skin-to-skin contact; breastfeeding; cesarean section; lactogenesis
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate SSC and early breastfeeding during CS group (Experimental): Receiving immediate SSC and early breastfeeding during CS and routine newborn care
  Interventions: Other: Immediate SSC and early breastfeeding during CS; Other: Routine newborn care
- control group (Other): Receiving delayed SSC and breastfeeding and routine newborn care
  Interventions: Other: Delayed SSC and breastfeeding after CS; Other: Routine newborn care

INTERVENTIONS:
Other: Immediate SSC and early breastfeeding during CS — Upon birth, the neonate is promptly placed prone on the mother's chest, with their head turned to one side for optimal skin contact. The drying process begins within 5 seconds and is completed within 20 to 30 seconds while the neonate remains on the mother's chest. Delayed cord clamping is practiced, with the cord clamped approximately 1-3 minutes after birth. Breastfeeding cues such as tongue movements or head turning are monitored, and the obstetric nurse assists the mother in initiating breastfeeding as soon as possible. SSC continues throughout the cesarean procedure, and upon completion, the newborn is temporarily separated from the mother for safety during transfer to the surgical cart. SSC is resumed immediately post-transfer and continues for a cumulative duration of at least 90 minutes. The neonate's skin color, breathing, and feeding responses are continuously observed.
  Arms: Immediate SSC and early breastfeeding during CS group
Other: Delayed SSC and breastfeeding after CS — The neonate is dried within 20-30 seconds after birth, the cord is clamped after 1-3 minutes, and then the neonate is sent to the ward to wait for the mother to complete the surgery. Immediate SSC is initiated within one hour after birth and maintained with the mother for at least 90 minutes post-surgery, during which the neonate's skin color and breathing are continuously monitored. The obstetric nurse supports the mother in initiating breastfeeding at the earliest opportunity.
  Arms: control group
Other: Routine newborn care — Newborn eye care, vitamin K1 administration, immunizations, weighing, and standard examinations are conducted before the neonate is transferred to the ward.

SUMMARY:
Background: Neonatal hypoglycemia is a prevalent and serious condition among late preterm and term infants, which can lead to severe neurodevelopmental consequences if not managed properly. Immediate skin-to-skin contact (SSC) and early initiation of breastfeeding are recognized as effective interventions to stabilize glucose levels and support neonatal adaptation to extrauterine life. However, implementing these practices during cesarean sections (CS) presents challenges due to the need to maintain a sterile surgical environment and logistical complexities.

Objective: This study aims to evaluate the effects of immediate SSC and early breastfeeding initiation during CS on neonatal hypoglycemia and breastfeeding outcomes.

Methods: A randomized controlled trial was conducted with 336 mother-neonate pairs undergoing elective CS. Participants were randomly assigned to either the experimental group, which received immediate SSC and early breastfeeding during CS, or the control group, which received standard care. Blood glucose levels of neonates were monitored at 1, 3, and 6 hours post-birth. Additional outcomes included the time to breastfeeding initiation, duration of the first breastfeeding session, onset of lactogenesis II, and the rate of exclusive breastfeeding during hospitalization.

DETAILED DESCRIPTION:
Neonatal hypoglycemia is a common condition among late preterm and term infants. It can lead to severe neurodevelopmental consequences if not managed properly. Immediate skin-to-skin contact (SSC) and early initiation of breastfeeding are effective interventions for stabilizing glucose levels and supporting neonatal adaptation to extrauterine life. While these practices are well-documented for their benefits in vaginal births, their implementation during cesarean sections (CS) presents challenges due to the need for maintaining a sterile surgical environment and the logistical complexities involved. The primary objective of this study was to evaluate the effects of immediate SSC and early breastfeeding initiation during CS on neonatal hypoglycemia and breastfeeding outcomes in late preterm and term infants.

This study was designed as a pragmatic, parallel-design, two-arm randomized controlled trial. It was conducted at Qingdao Municipal Hospital in China from July 2023 to July 2024. A total of 336 eligible mother-neonate pairs undergoing elective CS were included in the study.

Participants included mothers aged 18 years or older with a singleton pregnancy and gestational age between 34+1 and 41+6 weeks, undergoing elective CS with epidural or spinal anesthesia, willing to engage in SSC and breastfeeding during and after surgery, and newborns with Apgar scores above 8 at 1 and 5 minutes, a strong sucking reflex, and no critical conditions requiring transfer. Exclusion criteria involved serious pregnancy complications (e.g., placenta previa, eclampsia), conditions hindering SSC initiation (e.g., neonatal asphyxia, maternal excessive bleeding), and previous breast surgeries or medications affecting breastfeeding.

Participants were randomly assigned to either the experimental group (immediate SSC and early breastfeeding during CS) or the control group (standard care) using a block randomization sequence generated by Microsoft Excel 2010. The randomization process was centrally managed, with blinding maintained for staff performing SSC and data collectors, though patient blinding was not feasible.

Interventions:

Experimental Group:

1. SSC and Breastfeeding During CS: Immediately after delivery, the surgical drape was lowered for parents to witness the birth. The neonate was placed prone on the mother's chest and dried within 20-30 seconds. Breastfeeding was initiated as soon as possible, and SSC continued throughout the surgery and for at least 90 minutes post-transfer to the ward.
2. Routine Newborn Care: Included standard newborn care such as eye care, vitamin K1 administration, immunizations, and weighing, conducted before transferring the neonate to the ward.

Control Group:

1. Delayed SSC and Breastfeeding: SSC was initiated within one hour after birth and maintained for at least 90 minutes post-surgery. The neonate was dried within 20-30 seconds after birth and sent to the ward while the mother completed the surgery.
2. Routine Newborn Care: Similar to the experimental group.

Outcome Measures:

Primary Outcome: Incidence of neonatal hypoglycemia, with blood glucose levels monitored at 1, 3, and 6 hours post-birth using the Stat Strip Xpress glucose meter. Hypoglycemia was categorized as mild (<45 mg/dL), moderate-to-severe (<36 mg/dL), and severe (<18 mg/dL).

Secondary Outcomes: Included time to breastfeeding initiation, duration of the first breastfeeding session, onset of lactogenesis II (significant milk secretion perceived by the mother), and rate of exclusive breastfeeding during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* mothers aged 18 years or older with a singleton pregnancy, gestational age between 34+1 and 41+6 weeks.
* undergoing elective cesarean section with epidural, subarachnoid block, or combined spinal-epidural anesthesia, willing to engage in mother-infant SSC during and after the surgery, without experiencing severe reactions to anesthesia like vomiting or shivering that could affect SSC.
* having intention to breastfeed with no major contraindications (e.g., hepatitis B, syphilis, HIV, or other infectious diseases).
* newborns with Apgar scores above 8 at 1 and 5 minutes, a strong sucking reflex, and no critical neonatal conditions requiring transfer.

Exclusion Criteria:

* serious pregnancy complications such as placenta previa, placenta accreta spectrum, eclampsia, and grade 3 or higher cardiac issues per NYHA standards.
* challenges in initiating mother-infant SSC include emergencies such as neonatal asphyxia or respiratory distress, maternal excessive bleeding during surgery, and maternal infectious dermatoses.
* previous breast surgeries such as biopsies or augmentations, nipple inversions complicating breastfeeding, or taking medications affecting lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of neonatal hypoglycemia | 1, 3, and 6 hours after birth
  Neonatal blood glucose levels were assessed using the Stat Strip Xpress glucose meter at 1, 3, and 6 hours after birth. Hypoglycemia was categorized as follows: mild hypoglycemia (overall) at <45 mg/dL, moderate-to-severe at <36 mg/dL, and severe at <18 mg/dL. Treatment was initiated if levels dropped below 25 mg/dL or if symptoms like shakiness, tachycardia, pallor, hypothermia, hunger, sweating, or weakness appeared. In such cases, 10 ml/kg of formula was administered, followed by a recheck after 0.5 hour. If levels rise above 40 mg/dL, subsequent checks occurred every 3 hours. Persistent levels below 50 mg/dL necessitated continued formula feeding and monitoring, or transferred to neonatal care if needed.

SECONDARY OUTCOMES:
Breastfeeding initiation time | Assessment occurs immediately post-operation, with timing recorded to the minute.
  Characterized by newborns correctly latching onto the nipple and areola, and establishing regular, effective sucking and swallowing.
Duration of first breastfeeding | Assessment occurs immediately post-operation, with timing recorded to the minute.
  Start Timing at Latch-On: Begin timing when the infant first latches onto the breast.
  End Timing at Detachment: Stop timing when the infant detaches from the breast, either naturally or with assistance from the mother or healthcare provider.
Onset of lactogenesis II | The assessment occurs from surgery to pre-discharge, with timing recorded to the hour postpartum, an average of 72 hours.
  Marked by significant milk secretion perceived by the mother as breast fullness, confirmed by observing and squeezing the areola to assess milk spillage.
Exclusive breastfeeding rate during hospitalization | The assessment occurs from delivery to pre-discharge, an average of 5 days.
  This rate was calculated for mothers who underwent cesarean delivery in both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Qiao, Principal Investigator — Qingdao Municipal Hospital
Locations (1):
- Qingdao Municipal Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The paper needs to be submitted and published on a subscription basis, which has a longer cycle. Additionally, the data needs to be used for another paper, making it inconvenient to share.

REFERENCES:
- [Background] Cuschieri S. The CONSORT statement. Saudi J Anaesth. 2019 Apr;13(Suppl 1):S27-S30. doi: 10.4103/sja.SJA_559_18. PMID 30930716
- [Background] Wang X, Zhang X, Sobel HL, Li Z, Juan J, Yang H. Early essential newborn care for cesarean section newborns in China: study protocol for a multi-centered randomized controlled trial. Trials. 2022 Aug 19;23(1):696. doi: 10.1186/s13063-022-06615-z. PMID 35986372
- [Background] Roeper M, Hoermann H, Kummer S, Meissner T. Neonatal hypoglycemia: lack of evidence for a safe management. Front Endocrinol (Lausanne). 2023 Jun 8;14:1179102. doi: 10.3389/fendo.2023.1179102. eCollection 2023. PMID 37361517

DOCUMENTS (1):
  • Study Protocol (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT06543160/Prot_000.pdf